CLINICAL TRIAL: NCT06258993
Title: Increasing Physical Activity Among Breast Cancer Survivors: Use of the ORBIT Model to Refine and Test a Novel Approach to Exercise Promotion Based on Affect-regulation (Study 2)
Brief Title: A Randomized Two-Arm Proof of Concept Study Testing A Novel Approach to Exercise Promotion Based on Affect-regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Courtney J. Stevens, Assistant Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY02000934_2; K08CA259632 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affect-based Exercise Prescription (Affect-Rx) (Experimental)
  Interventions: Behavioral: Core Exercise Promotion Program; Behavioral: Affect-based exercise prescription
- Effort-based Exercise Prescription (RPE-Rx) (Active Comparator)
  Interventions: Behavioral: Core Exercise Promotion Program; Behavioral: Effort-based exercise prescription

INTERVENTIONS:
Behavioral: Core Exercise Promotion Program — Core intervention content will be delivered during the Visit 1 and 1-Month-Check-in meetings. Definitions of exercise will be provided, participants will be asked to discuss their past experiences with exercise, guidelines for being safe during exercise will be reviewed, and strategies for overcoming potential barriers to exercise will be discussed. All participants will be given an exercise plan organized according to the FIIT Principle (Frequency, Intensity, Time, and Type). The intensity component of the exercise plan will differ by study arm, all other elements will be delivered the same across both conditions. All participants will be given the goal of increasing weekly time spent exercising to ≥150 minutes, consistent with recommended guidelines. All participants will be given a smartwatch to support self-monitoring of exercise and activity levels throughout the 12-week study period.
Behavioral: Affect-based exercise prescription — Participants assigned to Affect-Rx will receive instructions to "select a pace of exercise that makes you feel as good as possible." The exercise intensity prescription section of their exercise plan will include the Feeling Scale as an attachment and participants will be given the instruction to "stay in the green zone" on the Feeling Scale.
  Arms: Affect-based Exercise Prescription (Affect-Rx)
Behavioral: Effort-based exercise prescription — Participants assigned to RPE-Rx will receive instructions to "select a pace that would make it challenging for you to carry on more than a short conversation." The exercise intensity prescription section of their exercise plan will include the Rating of Perceived Exertion (RPE) scale as an attachment and participants will be given the instruction to "stay in the green zone" on the RPE Scale.
  Arms: Effort-based Exercise Prescription (RPE-Rx)

SUMMARY:
The goal of this clinical trial is to test the effect of an affect-based exercise prescription on moderate-vigorous physical activity participation among survivors of breast cancer who completed primary treatment within the last 5 years. The main questions it aims to answer are:

1. Do at least 50% of participants assigned to the affect-based exercise prescription engage in ≥90 minutes of moderate-vigorous physical activity by the end of 12-weeks follow-up?
2. What level of satisfaction do breast cancer survivors who receive the affect-based exercise prescription report relative to breast cancer survivors who receive an effort-based exercise prescription.
3. What proportion of participants assigned to the affect-based exercise prescription stay enrolled in the study relative to the number of participants who stay enrolled in the effort-based exercise prescription.

All participants will:

* Be assigned to either the Affect-based exercise prescription or the Effort-based exercise prescription.
* Participate in two meetings with a member of the study team meant to help them get started increasing weekly exercise. These meetings are the same for all participants.
* Be asked to wear an activity monitor and respond to brief surveys for 10 straight days at 4 points in time: Baseline, 2weeks, 6weeks, and 12weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Within 5 years of completing primary cancer treatment (surgery, chemotherapy, and radiation) for Stage 0-III breast cancer
* <60 mins/week moderate-vigorous physical activity (MVPA) with no major changes for the past 6- months
* Own an Android or iPhone smartphone (or tablet) and willing to use it to complete app-based surveys during assessment periods
* Willing to wear the ActiGraph monitor during assessment periods
* Access to internet to complete REDCap survey assessments

Exclusion Criteria:

* Non-English speaking/not able to read English
* Evidence of major contraindications for exercise (informed by the 2020 Physical Activity Readiness-Questionnaire (PAR-Q)+)
* Currently pregnant
* History of severe mental illness or currently taking mood stabilizing medications (antipsychotics, anticonvulsants, or lithium)
* Evidence of moderate-severe depressive symptoms (indicated by a score≥ 10 on the Patient Health Questionnaire-8)
* Evidence of moderate-severe cognitive impairment (indicated by a score < 3 on a 6-item cognitive screener)
* Evidence of clinically significant substance use as indicated by a score of ≥ 2 on the CAGE- AID screener.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 2 Weeks Follow-up | 2-weeks follow-up assessment.
  The research grade ActiGraph wGT3X-BT model is a valid measure of physical activity intensity and duration among multiple populations, including breast cancer survivors. Minutes of moderate-vigorous physical activity will be collected from the ActiGraph wGT3X-BT every day for 10-days. Average minutes of moderate-vigorous physical activity completed per day of valid wear time will be calculated.
Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 6 Weeks Follow-up | 6-weeks follow-up assessment.
  The research grade ActiGraph wGT3X-BT model is a valid measure of physical activity intensity and duration among multiple populations, including breast cancer survivors. Minutes of moderate-vigorous physical activity will be collected from the ActiGraph wGT3X-BT every day for 10-days. Average minutes of moderate-vigorous physical activity completed per day of valid wear time will be calculated.
Average Minutes of Daily Moderate-vigorous Physical Activity Measured Using the ActiGraph wGT3X-BT Accelerometer at 12 Weeks Follow-up | 12-weeks follow-up assessment.
  The research grade ActiGraph wGT3X-BT model is a valid measure of physical activity intensity and duration among multiple populations, including breast cancer survivors. Minutes of moderate-vigorous physical activity will be collected from the ActiGraph wGT3X-BT every day for 10-days. Average minutes of moderate-vigorous physical activity completed per day of valid wear time will be calculated.

SECONDARY OUTCOMES:
Satisfaction With Study Participation as Measured by the Participant Satisfaction Questionnaire | 12-weeks follow-up assessment.
  An 8-item self-report questionnaire used to assess participant satisfaction with study participation using a Likert scale ranging from 1 to 4 . Scores are summed and then averaged; total scores range from 1- 4. Higher scores indicate greater satisfaction.
Study Retention at 2-weeks Follow-up | 2-weeks follow-up assessment.
  Number of participants who complete the 2-week follow-up assessment out of the number of participants who enroll in the study.
Study Retention at 6-weeks Follow-up | 6-weeks follow-up assessment.
  Number of participants who complete the 6-week follow-up assessment out of the number of participants who enroll in the study.
Study Retention at 12-weeks Follow-up | 12-weeks follow-up assessment.
  Number of participants who complete the 12-week follow-up assessment out of the number of participants who enroll in the study.
Acceptability of the Affect-regulated Exercise Prescription Measured Using the Treatment Acceptability and Preferences (TAP) Measure | 12-weeks follow-up assessment.
  A 4-item self-report questionnaire used to measure acceptability of the affect-regulated exercise prescription using a Likert scale ranging from 0 (not at all) to 4 (very much). Total scores range from 0 - 16. Higher scores indicate greater acceptability.
Change in Voluntary Exercise Behavior Measured Using The Voluntary Exercise Questionnaire | Baseline, 6-weeks follow-up, and 12-weeks follow-up.
  A 6-item self-report measure of exercise performed over the last month and week. Two items range from 1 (never) to 7 (often) and four items range from 0 (0 days per week) to 7 (7 days per week). Total scores range from 2-21. Higher scores reflect higher levels of voluntary exercise behavior.
Change in Physical Activity Category Completed in the Past Month Measured Using the Stanford Leisure-Time Activity Categorical Item (L-Cat) | Baseline, 6-weeks follow-up, and 12-weeks follow-up.
  A single item self-report measure that present six statements describing various levels of monthly physical activity. Response options range from 1 (I did not do much physical activity) to 6 (I did vigorous activities almost daily). Total scores range from 1-6. Higher scores reflect more vigorous, more frequent physical activities completed in the past month.
Change in Physical Activity using The International Physical Activity Questionnaire (IPAQ)-Short Form | Baseline, 6-weeks follow-up, and 12-weeks follow-up.
  A 7-item self-report measure calculating the amount of health-related vigorous and moderate-intensity physical activity as well as sitting time performed by adult participants over a one-week period. The number of minutes per day participants report for 3 categories vigorous, moderate, and walking activities are multiplied by the average metabolic equivalent (METs) for each category (8.0 METs, 4.9 METs, and 3.3 METs, respectively). Scores for each category are summed to calculate a physical activity score for the past week quantified as total MET values. Higher METS demonstrate a higher total volume of physical activity completed in the prior week. MET values between 0-599 are considered "low active," MET values between 600-1499 are considered "moderately active," and MET values 1500 or higher are considered "High active." This measure also assesses participants' total sitting time in the past week. Total number of minutes reported for sitting time is not part of the physical activity

OTHER OUTCOMES:
Change Overtime in Cancer-related Fatigue Measured Using the PROMIS Fatigue Short Form 8a | Baseline and 12-weeks follow-up assessments.
  An 8-item self-report measure with response options ranging from 1 (not at all) to 5 (very much) and fatigue interference ranging from 1 (never) to 5 (always) over the past 7 days. Total scores range from 8 - 40. Higher scores reflect more fatigue.
Change Overtime in Health-related Quality of Life Measured Using the PROMIS Global Health Scale | Baseline and 12-weeks follow-up assessments.
  A 10-item self-report measure with response options ranging from 1 (poor/never/not at all) to 5 (excellent/completely/always) for items 1-9 and 0 (no pain) to 10 (worst pain imaginable) for the item 10. Total scores range from 9 - 45. Higher scores represent better health-related quality of life.
Change Overtime in Physical Functioning Measured Using The PROMIS Physical Function Short Form 8a | Baseline and 12-weeks follow-up assessments.
  An 8-item self-report measure with response options ranging from 1 (unable to do) to 5 (without any difficulty) and the degree to which health limits specific activities on a scale from 1 (cannot do) to 5 (not at all). Total scores range from 8 - 40. Higher scores reflect better physical function.
Change Overtime in Anxiety measured using The PROMIS Anxiety Form | Baseline and 12-weeks follow-up assessments.
  An 8-item self-report measure with response options ranging from 1 (never) to 5 (always). Total scores range from 8 - 40. Higher scores reflect higher levels of anxiety.
Change Overtime in Depressive Symptoms using The PROMIS Depression Form | Baseline and 12-weeks follow-up assessments.
  An 8-item self-report measure with response options ranging from 1 (never) to 5 (always). Total scores range from 8 - 40. Higher scores reflect higher levels of depressive symptoms.
Change Overtime in Sleep Disturbance using The PROMIS Sleep Disturbance Scale | Baseline and 12-weeks follow-up assessments.
  An 8-item self-report measure with response options indicating the level of sleep disturbance a participant may experience. The first question asks about sleep quality and ranges from 1 (very good) to 5 (very poor). Questions 2-8 further inquire about the specifics of the sleep experience, ranging from 1 (not at all) to 5 (very much). Total scores range from 8 - 40. Higher scores reflect a greater degree of sleep disturbance or poorer quality of sleep.
Change Overtime in Intentions for Exercise Measured Using The Exercise Intentions Scale | Baseline, 6-weeks follow-up, and 12-weeks follow-up.
  A 5-item self-report measure of intentions to exercise in the next week. Response options range from 1 (not at all likely) to 7 (very likely). Responses are summed and then averaged; total scores range from 1-7. Higher scores represent stronger intentions to exercise in the next week.
Change Overtime in Physical Activity Enjoyment using the Physical Activity Enjoyment Scale-Short form (PACE-S) | Baseline, 6-weeks follow-up, and 12-weeks follow-up.
  A 4-item self-report measure with response options ranging from 1 (Strongly disagree) to 5 (Strongly agree). Total scores range from 4 - 20. Higher scores reflect higher levels of pleasure when performing physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney J Stevens, PhD, Principal Investigator — Dartmouth-Hitcock Health
Locations (1):
- Dartmouth-Hitchcock Clinic, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No